CLINICAL TRIAL: NCT03936907
Title: A Single-Dose, Randomized, Crossover Study to Compare the Safety, Tolerability and Pharmacokinetics of Medical Grade Cannabis - Orally Disintegrating Tablets (MGC-ODT) With Buccal Sativex®, in Healthy Adult Volunteers
Brief Title: Comparison of Safety, Tolerability and Pharmacokinetics of Medical Grade Cannabis (MGC) Orally Disintegrating Tablets With Buccal Sativex®, in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: One World Cannabis Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OWC-ODP12; 20185282 (Other: Israeli MOH)
Record Dates: First submitted 2019-02-12; First posted 2019-05-03 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-04

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — nabiximols

STUDY DESIGN:
Intervention Model Description: Sequence ABBA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orally Disintegrating MGC-ODT Tablet (Experimental): Administration of a single tablet of Medical Grade Cannabis - Orally Disintegrating Tablet (MGC-ODT) containing 5mg THC and 5 mg CBD
  Interventions: Drug: OWCP Orally Disintegrating Tablet
- Sativex® (Active Comparator): Sativex® spray X 2 actuations (1 under the tongue and 1 inside the cheek administered within 2 min) - Reference Product [Each 100 μL spray contains 2.7 mg THC and 2.5 mg CBD, total per administration: 5.4 mg THC and 5.0 mg CBD]
  Interventions: Drug: Sativex

INTERVENTIONS:
Drug: OWCP Orally Disintegrating Tablet — Medical Grade Cannabis - Orally Disintegrating Tablet (MGC-ODT) containing 5 mg THC and 5 mg CBD
  Arms: Orally Disintegrating MGC-ODT Tablet
Drug: Sativex — Sativex® Oromucosal Spray
  Arms: Sativex®

SUMMARY:
This is a preliminary study designed to assess the safety and properties of a new oral formulation containing the two most common cannabinoids used for medicinal purposes - Tetrahydrocannabinol (THC) and Cannabidiol (CBD). The formulation is designed to disintegrate sublingually in order to enhance absorption of these ingredients by circumventing first-pass metabolism by the liver (and probably also by the intestinal mucosal cells) as well as gastric acid degradation, thus allowing a rapid onset and more intensive pharmacological effect.

DETAILED DESCRIPTION:
This is a single-center, open-label, single-dose, crossover, randomized, pharmacokinetic study in healthy male adults.

Sixsteen (16) subjects will participate in the study. Each subject will undergo screening procedures within 28 days prior to dosing, to assess his eligibility to participate in the study.

Eligible subjects will participate in two dosing periods. They will be randomized to one of two administration sequences - AB or BA. In each period subjects will be admitted to the clinic on the evening before dosing. On the next morning, under fasting conditions they will receive one of the following administrations, according to a randomization list:

* Administration A: A single tablet of Medical Grade Cannabis - Orally Disintegrating Tablet (MGC-ODT) containing 5mg THC and 5 mg CBD (Test Formulation)
* Administration B: Sativex® spray X 2 actuations (1 under the tongue and 1 inside the cheek administered within 2 min) - Reference Product [Each 100 μL spray contains 2.7 mg THC and 2.5 mg CBD, total per administration: 5.4 mg THC and 5.0 mg CBD] A taste assessment questionnaire will be filled in by the subjects 2 minutes after drug administration (immediately following water administration).

Dosing will be followed by Pharmacokinetic (PK ) blood sampling for 24 hours and Adverse Events (AE) monitoring for the next 24 hours, at time points specified below.

A washout period of at least 2 weeks is required between the dosings.

An End-of Study (EOS)/Safety Follow-up visit will take place 7-10 days after the last dose of study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who provide written informed consent to participate in the study.
* Subjects who agree to have their name and details disclosed to the Israeli Ministry of Health and other responsible official authorities, as per the local legal requirement for participation in a THC study.
* Body Mass Index (BMI) ranging from 18 to <30 kg/m2.
* Subjects in general good health in the opinion of the investigator as determined by medical history, vital signs, ECG and a physical examination.
* No history of either recurrent or current buccal disorders (e.g. aphthae, xerostomia, infections).
* Supine blood pressure and heart rate within normal limits (systolic 90-140 mmHg; diastolic 50-90 mmHg, heart rate 45-100 beats per minute). No evidence of orthostatic hypotension.
* No clinically significant abnormalities in clinical laboratory parameters (hematology, blood chemistry, or urinalysis).
* Negative HIV 1/2, HBSAg, HCV serology tests at Screening.
* Subjects who agree to use an effective method of contraception during the course of the study. These include condom, having undergone a vasectomy or abstain from sexual intercourse.
* No known history of alcohol or drug abuse. Negative urinary screen for drugs of abuse as determined on the Screening visit and on admission before dosing.
* Willing to abstain from cannabis use 30 days before and throughout the study duration.
* Subjects must agree not to engage in potentially hazardous activities such as operating machinery, working at heights (e.g. maintenance and construction, climbing a ladder) throughout the study duration.
* Subjects must agree to abstain from driving from time of drug administration until 3 weeks after dosing.
* Subjects must agree to eat all the food and beverages provided during the study, and only these meals.
* Subjects must be able to understand the requirements of the study and must be willing to comply with the requirements of the study.

Exclusion Criteria:

* Known history of significant medical disorders including: cardiac, gastroenterological, hepatic, renal, endocrine, neurological, hematological, neoplastic, immunological, skeletal (or other) that, as per the medical judgment of the principal investigator, could interfere with the execution and/or results of the study or contraindicates administration of the study medications.
* History of fainting or recurrent dizziness.
* History of epilepsy/seizures.
* History of any significant psychiatric disorder i.e., mania, depression, or schizophrenia.
* Any known or suspected history or family history of schizophrenia, or other psychotic illness, history of severe personality disorder or other severe significant psychiatric disorder other than reactive depression.
* Known hypersensitivity to cannabinoids (including cannabis extracts), excipients of tablet or of Sativex.
* Any history of cannabis dependence.
* Any history of adverse events associated with cannabis intoxication.
* A history of drug or alcohol abuse, or a history of regular alcohol consumption (by declaration) within 6 months of the study, defined as an average weekly intake of >14 drinks. One drink is equivalent to 12 grams of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.

Positive urine drug of abuse test on Screening and on admission to the CRC before dosing.

* A positive alcohol breath test on admission to the CRC before dosing.
* History of clinically significant drug allergy; history of atopic allergy (asthma, urticaria, eczematous dermatitis).
* Any clinically significant abnormality upon physical examination or in the clinical laboratory tests at the Screening visit.
* Liver disease or liver injury manifested by clinically significant abnormal liver function tests
* Subjects receiving concomitant antipsychotic, sedative, hypnotic or other psychoactive drugs.
* Use of any prescription or over-the-counter (OTC) medications, vitamins and herbal or dietary supplements including St. John's Wort within 14 days prior to anticipated dosing; subjects who had treatment with any known enzyme-altering agent (e.g. CYP3A4 inducers or inhibitors), within 30 days of dosing. Paracetamol for symptomatic relief of pain is allowed until 24 hours prior to study drug administration.
* Any acute illness (e.g. acute infection) within 72 hours prior to study drug administration that is considered of significance by the Principal Investigator.
* Oral piercing of the tongue, inner lip or cheek.
* Presence of mouth ulcerations or any abnormalities of the oral cavity.
* Unwilling to abstain from smoking throughout the in-house stay at the CRC.
* Unwilling to abstain from alcohol use throughout the in-house stay at the CRC.
* Subjects who refuse to avoid strenuous physical activity throughout in-house stay in the CRC.
* Participation in another clinical trial with drugs received within 3 months prior to first dosing (calculated from the previous study's last dosing date).
* Subjects who donated blood in the 3 months or received blood or plasma derivatives in the 6 months preceding study drug administration.
* Subjects with an inability to communicate well with the investigators and CRC staff (i.e., language problem, poor mental development or impaired cerebral function).
* Inability to fast or consume the food provided in the study (including any known food allergies or food restrictions such as lactose intolerance or gluten-free diet).
* Subjects who are non-cooperative or unwilling to attend scheduled clinic visits and/or comply with the study protocol.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-07-18 (Actual); Study Completion 2019-07-18 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter- Tmax determined from plasma concentrations of THC, 11-hydroxy-THC and CBD. | 24 hours post dosing
  he amount of time requires for THC, 11-hydroxy-THC and CBD to reach to maximum concentration in serum
Pharmacokinetic parameter -Cmax determined from plasma concentrations of THC, 11-hydroxy-THC and CBD. | 24 hours post dosing
  Mean highest observed plasma concentration of THC, 11-hydroxy-THC and CBD after dosing.
Pharmacokinetic parameter- AUC0-t (area under the plasma concentration-time curve) determined from plasma concentrations of THC, 11-hydroxy-THC and CBD. | 24 hours post dosing
Pharmacokinetic parameter- T½ determined from plasma concentrations of THC, 11-hydroxy-THC and CBD. | 24 hours post dosing
  The time required for the concentration of THC, 11-hydroxy-THC and CBD to reach half of its original value
Pharmacokinetic parameter- kel determined from plasma concentrations of THC, 11-hydroxy-THC and CBD. | 24 hours post dosing
  Elimination rate constant K - The rate at which THC, 11-hydroxy-THC and CBD are removed from the body determined by their plasma concentration.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerabilityof MGC-ODTand Sativex® ] | 2 weeks post dosing
  Safety

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel (isr), Israel

IPD SHARING:
Plan to Share IPD: No